# RESEARCH STUDY INFORMATION SHEET

Study to be Conducted at: Greenville Memorial Hospital

701 Grove Road Greenville, SC 29605

Study Sponsor: Greenville Health System and Clemson University

Principal Investigator: Steve Lowe, MD

#### INTRODUCTION

You are being asked to participate in a research study. The Institutional Review Board of the Greenville Health System has reviewed this study for the protection of the rights of human participants in research studies, in accordance with federal and state regulations. However, before you choose to be a research participant, it is important that you read the following information and ask as many questions as necessary to be sure that you understand what your participation will involve.

## **PURPOSE AND PROCEDURES**

You are being asked to participate in this study to further our understanding of factors influencing how physicians order imaging tests.

We plan to enroll 150-200 participants in this study. Your participation will involve a short computer simulation (estimated 5-10 minutes to complete) featuring clinical vignettes and clinical decision making.

## **POSSIBLE RISKS AND BENEFITS**

There are no known medical risks related to participation in this study. The greatest risk is the possible release of your personal information. Your study records are considered confidential, but absolute confidentiality cannot be guaranteed. This study may result in presentations and publications, but steps will be taken to make sure you are not identified by name. The possible benefits are educational in nature, including exposure to evidence based medicine data, cost data related to the patient experience, and relevant legal case law having to do with Head CT scans.

### **VOLUNTARY PARTICIPATION**

Participation in this study is completely voluntary. You may refuse to participate or withdraw from the study at any time. If you refuse to participate or withdraw from the study, you will not be penalized or lose any benefits. Your decision will not affect your relationship with the investigators or the Greenville Health System.

#### **CONTACT FOR QUESTIONS**

For more information concerning this study and research-related risks or injuries, or to give comments or express concerns or complaints, you may contact the study co-investigator Zachary A. Connor, MD by email at <a href="mailto:zconnor@ghs.org">zconnor@ghs.org</a> or by phone at 978-944-2899. You may also contact a representative of the Institutional Review Board of the Greenville Health System for information regarding your rights as a participant involved in a research study or to give comments or express concerns, complaints or offer input. You may obtain the name and number of this person by calling (864) 455-8997. A survey about your experience with this informed consent process is located at the following website:

https://www.surveymonkey.com/s/T5C86P8

Participation in the survey is completely anonymous and voluntary and will not affect your relationship with the Greenville Health System. If you would like to have a paper copy of this survey, please tell the principal investigator.

Greenville Health System
IRB Number: Pro00054122
Approved: 5/25/2016